CLINICAL TRIAL: NCT04235452
Title: Electrophysiological Characteristics and Anatomical Differentiation of Epileptic and Non-epileptic Myoclonus.
Status: Completed | Type: Observational
Sponsor: Mansoura University Hospital (Other)
Responsible Party: Principal Investigator, Ahmed Esmael, Assistant Prof of Neurology, Mansoura University Hospital
Other Study IDs: Mansoura University 11
Record Dates: First submitted 2020-01-16; First posted 2020-01-22 (Actual); Last update posted 2020-01-22 (Actual); Status verified 2020-01

CONDITIONS: Myoclonus; Evoked Potential
Keywords: Myoclonus, Evoked potential
MeSH Terms: conditions — Myoclonus | interventions — Evoked Potentials, Somatosensory

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Epileptic myoclonus: Juvenile Myoclonic Epilepsy and Progressive Myoclonic Epilepsy
  Interventions: Diagnostic Test: Somatosensory evoked potential
- Non-epileptic myoclonus (secondary): Post hypoxic myoclonus, Post ischemic stroke myoclonus, Hepatic, Chronic kidney disease, and Drug induced myoclonus
  Interventions: Diagnostic Test: Somatosensory evoked potential

INTERVENTIONS:
Diagnostic Test: Somatosensory evoked potential — Stimulation of the right and left median nerves for each subject were carried out with electrical square wave pulses of 0.2 ms duration applied at a rate of 5 HZ. with cathode proximally. The intensity of the stimulus was adjusted to produce minimal twitches of the thumb (1-2 cm thumb movement). Five hundred (500) stimuli were delivered. The recording electrode picked up the responses. They were then summated and averaged.
  The final evoked potential was then displayed on the screen. When two reproducible SEPs responses were obtained the data was accepted for analysis. The graph was printed out on paper, for the purpose of simplification only one response was printed out.

SUMMARY:
This study was conducted on a series of patients with myoclonus to identify the electrophysiological characteristics and the anatomical classification of myoclonus of different causes.

DETAILED DESCRIPTION:
The current study included 50 patients with different types of myoclonus in comparison to 30 control subjects. Electrophysiological study was done for all patients by Somatosensory Evoked Potential (SSEP) and Electroencephalography (EEG) while the control group underwent SSEP. SSEP was studied in the patients and control group by stimulation of right and left median nerves.

ELIGIBILITY:
Inclusion Criteria:

* Myoclonus classified into primary and secondary myoclonus.

Exclusion Criteria:

* Psychiatric comorbidity to exclude psychological myoclonus.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: 50 patients with myoclonus of different etiologies (primary and secondary myoclonus).
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2019-08-31 (Actual); Study Completion 2019-10-31 (Actual)

PRIMARY OUTCOMES:
Somatosensory evoked potential | 24-72 hours
  Stimulation of the right and left median nerves for each subject were carried out with electrical square wave pulses of 0.2 ms duration applied at a rate of 5 HZ. with cathode proximally. The intensity of the stimulus was adjusted to produce minimal twitches of the thumb (1-2 cm thumb movement). Five hundred (500) stimuli were delivered. The recording electrode picked up the responses. They were then summated and averaged.
  The final evoked potential was then displayed on the screen. When two reproducible SEPs responses were obtained the data was accepted for analysis. The graph was printed out on paper, for the purpose of simplification only one response was printed out.

CONTACTS AND LOCATIONS:
Overall Officials: Esmael Ahmed, MD, Principal Investigator — Assistant Prof of Neurology
Locations (1):
- Mansoura University Hospital, Al Mansurah, Dakahlia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Abdo WF, van de Warrenburg BP, Burn DJ, Quinn NP, Bloem BR. The clinical approach to movement disorders. Nat Rev Neurol. 2010 Jan;6(1):29-37. doi: 10.1038/nrneurol.2009.196. PMID 20057497
- [Result] Agarwal P, Frucht SJ. Myoclonus. Curr Opin Neurol. 2003 Aug;16(4):515-21. doi: 10.1097/01.wco.0000084231.82329.9c. PMID 12869812
- [Result] Alvarez, V. & Rossetti, A. O. 2015. Electroencephalography and Evoked Potentials: Technical Background. Clinical Neurophysiology in Disorders of Consciousness. Springer. 7-23.